CLINICAL TRIAL: NCT00502060
Title: A Phase I Open-Label Study to Assess the Safety, Tolerability and PK of Ascending Multiple Oral Doses of AZD2171 When co-Administered With Fixed Multiple Oral Doses of ZD1839 (250mg or 500mg Once Daily) in Patients With Advanced Cancer
Brief Title: Phase I Study of AZD2171 co-Administered With Fixed Multiple Oral Doses of ZD1839 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00004
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Advanced Tumor
Keywords: Phase I; AZD2171; ZD1839; solid tumor
MeSH Terms: interventions — cediranib; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AZD2171
Drug: ZD1839

SUMMARY:
Phase I AZD2171 in combination with ZD1839 study recruiting patients with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* tumor progressed on standard therapy or ineligible for standard therapy
* life expectancy of 12 weeks or more
* WHO performance status 0-2

Exclusion Criteria:

* History of active interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2004-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
primary objective is to determine the safety and tolerability of multiple oral doses fo AZD2171 when co-administered with fixed daily oral doses of ZD1839

SECONDARY OUTCOMES:
to explore the PK of AZD2171 when given alone for 7 days and in combination with ZD1839 for 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Nick Botwood, BSc, MBBS, MRCP, MFPM, Study Director — AstraZeneca; G Giaccone, Prof, Principal Investigator — Vrije Universiteit Medical Centre
Locations (3):
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
  - Research Site, Utrecht